CLINICAL TRIAL: NCT01723566
Title: Panorama 2 Medtronic CRDM Implantable Cardiac Device Long Term Registry
Brief Title: PANORAMA 2 Observational Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: PANORAMA 2
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-08

CONDITIONS: Heart Rhythm Disorders
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Understanding the clinical practice of treatment of cardiac rhythm disorders all over the world and understanding the clinical outcomes of the treatment with its cardiac rhythm products in real world patient population is essential for Medtronic to be able to effectively develop new products and adjust existing products. In addition Medtronic is committed to monitor the safety of its products throughout the entire life cycle to ensure maximum product reliability.

The Panorama 2 registry will enable Medtronic to increase data collection of clinical practice with Medtronic implantable Cardiac Rhythm and Disease Management (CRDM) devices in various regions across the world and on product reliability of its CRDM devices.

ELIGIBILITY:
Inclusion criteria:

* Patient is 18 years of age or older (lower age limit dependent on local law: to be specified in country-specific addendum to the clinical investigational plan, if applicable)
* Patient or Legally Authorized Representative provides signed and dated authorization and/or consent per institution and local requirements
* Patient will be treated with a commercially available implantable Medtronic CRDM device/ Vitatron device within maximally 30 days after enrollment or within 3 days prior to enrollment

Exclusion criterion:

• Patient has exclusion criteria per local law (to be specified in country-specific addendum to the clinical investigational plan, if applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that have a Medtronic implantable CRDM Device implanted (including Vitatron), which is commercially available at the start of the registry or becomes commercially available during the course of the registry, and used within its intended use, may be included.
  These products are:
  * Pacemaker systems: Implantable Pulse Generators (IPG) and cardiac leads
  * Defibrillation systems: Implantable Cardioverter Defibrillators (ICD) and cardiac leads
  * Resynchronization systems: Cardiac Resynchronization Therapy (CRT):
    * Cardiac Resynchronization Therapy - Pacemaker (CRT-P) and cardiac leads
    * Cardiac Resynchronization Therapy - Defibrillator (CRT-D) and cardiac leads
  * Implantable Loop Recorders (ILR)
Sampling Method: Non-Probability Sample
Enrollment: 4706 (Actual)
Dates: Start 2012-07-25 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

PRIMARY OUTCOMES:
Describe region-specific clinical practice of CRDM device use | 2012-2019
  To describe the region-specific current clinical practices associated with the device treatment of patients receiving implantable Medtronic CRDM devices by collecting information on the patient characteristics (demographics, medical history and cardiovascular status), the type of Medtronic CRDM devices used, the indication for the use of the Medtronic CRDM devices and the clinical outcomes of the treatment with the Medtronic CRDM devices (all deaths, cardiovascular hospitalizations, Serious Adverse Device Effects and NYHA class).

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospital, Cairo, Egypt